CLINICAL TRIAL: NCT06218550
Title: The Effect of Delta-8-THC vs Delta-9-THC on Simulated Driving Performance and Measures of Impairment
Brief Title: Delta-8-THC vs. Delta-9-THC on Simulated Driving Performance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00394164
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; delta-8-tetrahydrocannabinol

STUDY DESIGN:
Intervention Model Description: A within-subjects design. At the time of study randomization, participants will be assigned to complete Sub-Study 1 followed by Sub-Study 2, or vice versa, using a counter-balanced randomization sequence. The order in which dose conditions are administered within each sub-study will be randomized across participants because there are too many drug conditions to fully counterbalance dosing within sub-studies at the proposed sample size.
Who Masked: Participant, Outcomes Assessor
Masking Description: Placebo controlled, double blind drug administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Oral Placebo (Placebo Comparator): A brownie containing no experimental drugs will be eaten by study participants
  Interventions: Drug: Placebo
- Oral administration of 30mg ∆8-THC (Experimental): A brownie infused with 30mg ∆8-THC will be eaten by study participants
  Interventions: Drug: Delta-8-THC
- Oral administration of 60mg ∆8-THC (Experimental): A brownie infused with 60mg ∆8-THC will be eaten by study participants
  Interventions: Drug: Delta-8-THC
- Oral administration of 30mg ∆9-THC (Experimental): A brownie infused with 30mg ∆9-THC will be eaten by study participants
  Interventions: Drug: Delta-9-THC
- Administration of vaporized Placebo (Placebo Comparator): Participants will inhale ambient air through a handheld vaporizer (minimum 15 "puffs")
  Interventions: Drug: Placebo
- Administration of vaporized 30mg ∆8-THC (Experimental): Participants will inhale 30mg ∆8-THC using a handheld vaporizer (minimum 15 "puffs")
  Interventions: Drug: Delta-8-THC
- Administration of vaporized 60mg ∆8-THC (Experimental): Participants will inhale 60mg ∆8-THC using a handheld vaporizer (minimum 15 "puffs")
  Interventions: Drug: Delta-8-THC
- Administration of vaporized 30mg ∆9-THC (Experimental): Participants will inhale 30mg ∆9-THC using a handheld vaporizer (minimum 15 "puffs")
  Interventions: Drug: Delta-9-THC

INTERVENTIONS:
Drug: Delta-9-THC — Acute self-administration of inhaled or oral ∆9-THC by healthy adult research volunteers
  Arms: Administration of vaporized 30mg ∆9-THC; Oral administration of 30mg ∆9-THC
Drug: Delta-8-THC — Acute self-administration of inhaled or oral ∆8-THC by healthy adult research volunteers
  Arms: Administration of vaporized 30mg ∆8-THC; Administration of vaporized 60mg ∆8-THC; Oral administration of 30mg ∆8-THC; Oral administration of 60mg ∆8-THC
Drug: Placebo — Consumption of a brownie or inhalation of ambient air through a cannabis vaporizer by health adult research volunteers
  Arms: Administration of vaporized Placebo; Oral Placebo

SUMMARY:
Delta-8-THC is an isomer of delta-9-THC that has become widely available due to the legalization of hemp and its derivatives. Very little controlled research has been conducted with delta-8-THC and some research suggests it produces similar effects to delta-9-THC, albeit at lower potency. The present study will evaluate the dose effects of delta-8-THC, compared with delta-9-THC, on simulated driving performance, field sobriety tests, cognitive performance, and biomarkers of exposure to cannabinoids. The results will inform policy and education related to impairment due to acute delta-8-THC exposure via vaporization and oral ingestion.

DETAILED DESCRIPTION:
The present study will characterize the acute effects of oral and inhaled ∆8-THC, compared with a positive control dose of ∆9-THC and placebo, on subjective drug effects, cardiovascular effects, cognitive performance, simulated driving performance, field sobriety tests, and drug testing outcomes in oral fluid, blood, hair, and urine. Healthy adults with a history of cannabis use will be recruited to participate in a placebo-controlled, within-subject crossover study at the Johns Hopkins Behavioral Pharmacology Research Unit (BPRU). The result will be a comparative pharmacology and toxicology dataset for ∆8-THC and ∆9-THC via both oral ingestion and inhalation, two routes of administration that are predominant in retail products currently being sold across the U.S. This study will provide urgently needed data on the behavioral pharmacology and toxicology of ∆8-THC, a novel cannabinoid that is now widely available, but for which there is little public knowledge or public health messaging. This data will directly inform the impact of ∆8-THC use on drug testing programs, and the comparative effects of ∆8-THC to ∆9-THC can be used to inform regulatory decisions related to public safety and the sale of these products.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 55
2. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
3. Test negative for recent cannabis use prior to each experimental test session
4. Test negative for drugs of abuse and alcohol prior to each experimental test session
5. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission
6. Have a body mass index (BMI) in the range of 19 to 36 kg/m2
7. Report use of cannabis in the past 3 years (both sub-studies) and prior experience inhaling cannabis (either via smoking or vaporization) for vaporization sub-study participation
8. Have not donated blood in the prior 30 days.
9. Have a current government-issued driver's license

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than nicotine, alcohol, or caffeine in the month prior to study participation.
2. History of or current evidence of health issues judged by the investigator to put the participant at greater risk of experiencing an adverse event due to drug exposure or completion of other study procedures.
3. Current concomitant medication use that may interact with the study drug (∆8-THC and ∆9-THC).
4. History of xerostomia (dry mouth), or the presence of mucositis, gum infection or bleeding, or other significant oral cavity disease or disorder that in the investigator's opinion may affect the collection of oral fluid samples.
5. Participation in other research projects that could impact the present study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) in cm | 0-8 hours
  A measure of lane weaving during simulated driving performance, the standard deviation of lateral position is a standard metric of impairment in driving performance. A score of 0 (perfect score, no deviation) is the minimum score possible and there is no upper threshold score. Higher scores equate to worse performance (more lane weaving).

SECONDARY OUTCOMES:
Mean Peak Change From Baseline Drug Effect Rating as Assessed by the Drug Effect Questionnaire (DEQ) | 0-8 hours
  Peak rating (0-100) of Drug Effect on the DEQ, a visual analog scale (VAS) self-report questionnaire with 0 being No drug effect and 100 being maximum drug effect
Mean Peak Change From Baseline Global Impairment Score as assessed by the DRiving Under the Influence of Drugs (DRUID) App | 0-8 hours
  Peak Global Impairment score (0-75) recorded as a result of performance on the DRUID App, a brief cognitive task battery completed on a mobile device (e.g., iPad). Larger scores indicate worse performance on the task.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No